CLINICAL TRIAL: NCT05586555
Title: A Monocentric Study Evaluating Pupillometry as an Objective Measurement for Cochlear Implant (CI) Fittings
Brief Title: A Monocentric Study Evaluating Pupillometry as an Objective Measurement for CI Fittings
Acronym: PupillOM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Demant's transfer of its cochlear implant activity to Cochlear. Slow recruitment and misalignment with Cochlear's interests are also determining factors.
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OM29
Record Dates: First submitted 2022-09-20; First posted 2022-10-19 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss, Bilateral; Cochlear Hearing Loss; Hearing Loss, Cochlear
Keywords: Cochlear Implant system
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Bilateral

STUDY DESIGN:
Intervention Model Description: A control group with normal hearing subjects versus a CI group with cochlear implanted subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (normal hearing in regards of age) (Other): Normal hearing participants according to pure tone hearing levels defined for age and tested frequency (audiometry ISO 7029 and Wang & Puel, 2020 recommendations for hearing loss at the tested frequencies). Total of 32 subjects in this arm.
  Interventions: Other: Pupillometry (Eve-tracking measurements)
- CI group (cochlear implanted subjects) (Experimental): Cochlear implanted subjects with bilateral, severe-to-profound sensorineural hearing loss, with at least one Oticon Medical cochlear implant system .
  Up to 40 subjects in this arm:
  * 20 subjects will perform experiment 1 & 2
  * 20 subjects will perform experiment 3
    * The subjects of the experiment 3 ore either those taken part to experiment 1 and 2, or subjects who only take port to the experiment 3
  Interventions: Other: Pupillometry (Eve-tracking measurements)

INTERVENTIONS:
Other: Pupillometry (Eve-tracking measurements) — Pupillometry measurements are carried out by a dedicated device (eye tracker), which includes cameras allowing the measurement of pupillary dilation. The subject stands in front of a screen and fixes a point in the center of the screen, the cameras placed on the screen allowing a measurement of the pupillary dilation in a non-invasive way. These eye-tracking measurements are performed simultaneously with an auditory task and allow to study the pupil's response to different stimuli.

SUMMARY:
This trial is a monocentric, prospective and controlled study of the pupil response to detect hearing threshold and comfortable loudness of normal-hearing (NH) and CI-subjects.

DETAILED DESCRIPTION:
The purpose of the clinical investigation is to explore the pupil dilation response of subjects with a cochlear implant and to provide proof of concept that it is possible to perform the adaptation of a cochlear implant using pupillometry.

The population of this study is divided in 2 group:

* A control group with normal-hearing listeners.
* An Cl group with subjects with bilateral, severe-to-profound sensorineural hearing loss, with at least one cochlear implant for more than 6 months.

Mainly used in audiology to evaluate listening effort, pupillometry is an objective measure that could also be used for fittings. Studies have shown that sound intensity influence pupil dilation. indeed, normal hearing and hearing aids subjects exhibit larger pupil responses with increasing intensity/loudness. The purpose of this study is to explore the pupil dilation response of cochlear implant subjects and to provide a proof of concept that we can perform cochlear implant fitting using pupillometry.

Implanted subjects (Cl group) will undergo up to 3 visits:

1. Visit 1 or V1(inclusion) on day 1,
2. Visit 2 or V2 (Experiment 1-+2+3 or Experiment 1+2 or Experiment 3 )* up to 1 month after V1
3. Visit 3 or V3 (Experiment 1+2 or Experiment 3, optional)* up to 1 month after V2 *lt is up to investigator decision to conduct experiment 1+2 and experiment 3 the same day or in on independent visit (no matter in which order)

Normal-hearing listeners (control group) will undergo up to 2 visits:

1. Visit 1 or Va (inclusion) on day 1,
2. Visit 2 or V2 (experiment) up to 1 month after V1

ELIGIBILITY:
Inclusion Criteria:

* Both groups:

  * Adult (≥ 18 years old)
  * Fluent in French language
  * Affiliation to social security
  * Information and signature of a written consent prior to any study-specific procedure
* Control group (normal hearing in regards of age):

  • Normal hearing participants according to pure tone hearing levels defined for age and tested frequency (audiometry ISO 7029 and Wand & Puel, 2020 recommendations for hearing loss at the tested frequencies)
* CI group (cochlear implant subjects):

  * Bilateral, severe-to-profound sensorineural hearing loss, with at least one cochlear implant system
  * Using Oticon Medical Neuro Cochlear Implant System (NCIS) or Digisonic Cochlear Implant system (DCIS), unilateral or bilateral
  * Duration of cochlear implant experience ≥ 6 months (period from cochlear implant activation to study enrolment)
  * Pure Tone Audiometry must be strictly below 50 dBA, CI aided.

Exclusion Criteria:

* Both groups, according to the best practices for pupillometry (Winn et al., 2018):

  * Eye diseases: nystagmus, amblyopia, and macular degeneration
  * Severe head injury or any history of significant neurological problems: These issues can affect gaze stability, congruence of eye movements, and pupil dilation
  * Concomitant medication that can impact the parasympathetic autonomic nervous system
  * Person under State Medical Assistance (AME for "Aide medical d'état" in French)
  * Use of one of the following treatments: Trihexyphenidyl, Biperiden or Tropatepine (anticholinergics, commonly used in the treatment of Parkinson's disease)
  * Person under legal protection (guardianship, curators, other, etc.) or under family authorization
  * Unwillingness or inability to comply with all investigational requirements
  * Additional cognitive, medical, or social handicaps that would prevent completion of all study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Measurement of the pupil dilation response to a range of auditory stimuli (acoustic and electric). | At Visit 2 (Month 1)
  Pupil dilation response for each intensity and frequency [Mean pupil dilatation in milimeters]

SECONDARY OUTCOMES:
Evaluation of the loudness perception of the subjects regarding the different auditory stimuli (acoustic and electric) to correlate the results to the pupil dilation response. | At Visit 2 (Month 1) and Visit 3 (Month 2)* [* if done]
  Loudness score corresponding to each pupil dilation response. [Using Oticon Medical Loudness scale: scale from 0 to 10 following the ISO 16832. 0 (zero) corresponding to inaudible level and 10 to extremely loud (intolerable) sounds.]

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Mosnier, Principal Investigator — Centre de Recherche en Audiologie adulte - CreA- GH Pitié Salpêtrière (APHP)
Locations (1):
- Centre de Recherche en Audiologie adulte GH Pitié-Salpêtrière, APHP Sorbonne Université, Unité Fonctionnelle Implants auditifs et Explorations Fonctionnelles, 52 Bd Vincent Auriol, 75013 Paris, France, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang J, Puel JL. Presbycusis: An Update on Cochlear Mechanisms and Therapies. J Clin Med. 2020 Jan 14;9(1):218. doi: 10.3390/jcm9010218. PMID 31947524
- [Background] Vaerenberg B, Smits C, De Ceulaer G, Zir E, Harman S, Jaspers N, Tam Y, Dillon M, Wesarg T, Martin-Bonniot D, Gartner L, Cozma S, Kosaner J, Prentiss S, Sasidharan P, Briaire JJ, Bradley J, Debruyne J, Hollow R, Patadia R, Mens L, Veekmans K, Greisiger R, Harboun-Cohen E, Borel S, Tavora-Vieira D, Mancini P, Cullington H, Ng AH, Walkowiak A, Shapiro WH, Govaerts PJ. Cochlear implant programming: a global survey on the state of the art. ScientificWorldJournal. 2014 Feb 4;2014:501738. doi: 10.1155/2014/501738. eCollection 2014. PMID 24688394
- [Background] Legris E, Galvin J, Mofid Y, Aguillon-Hernandez N, Roux S, Aoustin JM, Gomot M, Bakhos D. Relationship between Behavioral and Objective Measures of Sound Intensity in Normal-Hearing Listeners and Hearing-Aid Users: A Pilot Study. Brain Sci. 2022 Mar 15;12(3):392. doi: 10.3390/brainsci12030392. PMID 35326347
- [Background] Versfeld NJ, Lie S, Kramer SE, Zekveld AA. Informational masking with speech-on-speech intelligibility: Pupil response and time-course of learning. J Acoust Soc Am. 2021 Apr;149(4):2353. doi: 10.1121/10.0003952. PMID 33940918
- [Background] Dingemanse G, Goedegebure A. Listening Effort in Cochlear Implant Users: The Effect of Speech Intelligibility, Noise Reduction Processing, and Working Memory Capacity on the Pupil Dilation Response. J Speech Lang Hear Res. 2022 Jan 12;65(1):392-404. doi: 10.1044/2021_JSLHR-21-00230. Epub 2021 Dec 13. PMID 34898265
- [Background] Bala ADS, Whitchurch EA, Takahashi TT. Human Auditory Detection and Discrimination Measured with the Pupil Dilation Response. J Assoc Res Otolaryngol. 2020 Feb;21(1):43-59. doi: 10.1007/s10162-019-00739-x. Epub 2019 Dec 2. PMID 31792632
- [Background] Jackson IR, Sirois S. But that's possible! Infants, pupils, and impossible events. Infant Behav Dev. 2022 May;67:101710. doi: 10.1016/j.infbeh.2022.101710. Epub 2022 Mar 17. PMID 35306326
- [Background] Kaldy Z, Blaser E. Putting effort into infant cognition. Curr Dir Psychol Sci. 2020 Apr;29(2):180-185. doi: 10.1177/0963721420903015. Epub 2020 Feb 27. PMID 33746375
- [Background] Russo FY, Hoen M, Karoui C, Demarcy T, Ardoint M, Tuset MP, De Seta D, Sterkers O, Lahlou G, Mosnier I. Pupillometry Assessment of Speech Recognition and Listening Experience in Adult Cochlear Implant Patients. Front Neurosci. 2020 Nov 6;14:556675. doi: 10.3389/fnins.2020.556675. eCollection 2020. PMID 33240035
- [Background] Schramm D, Chen J, Morris DP, Shoman N, Philippon D, Caye-Thomasen P, Hoen M, Karoui C, Laplante-Levesque A, Gnansia D. Clinical efficiency and safety of the oticon medical neuro cochlear implant system: a multicenter prospective longitudinal study. Expert Rev Med Devices. 2020 Sep;17(9):959-967. doi: 10.1080/17434440.2020.1814741. Epub 2020 Oct 3. PMID 32885711
- [Background] Sulas E, Hasan PY, Zhang Y, Patou F. Streamlining experiment design in cognitive hearing science using OpenSesame. Behav Res Methods. 2023 Jun;55(4):1965-1979. doi: 10.3758/s13428-022-01886-5. Epub 2022 Jul 6. PMID 35794416
- [Background] Winn MB, Wendt D, Koelewijn T, Kuchinsky SE. Best Practices and Advice for Using Pupillometry to Measure Listening Effort: An Introduction for Those Who Want to Get Started. Trends Hear. 2018 Jan-Dec;22:2331216518800869. doi: 10.1177/2331216518800869. PMID 30261825